CLINICAL TRIAL: NCT04990375
Title: Placebo-controlled Randomized Clinical Trial: tDCS to Prevent Relapse in Alcohol Use Disorder
Brief Title: tDCS to Prevent Relapse in Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Macha Dubuson, Principal Investigator, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tDCS in AUD
Record Dates: First submitted 2021-07-13; First posted 2021-08-04 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Active tDCS; Sham tDCS
Keywords: tDCS; DLPFC; Alcohol use disorder; Relapse; Craving
MeSH Terms: conditions — Alcoholism; Recurrence | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: active tDCS vs. sham tDCS, while the patient is watching a documentary
Who Masked: Participant
Masking Description: sham tDCS protocol: 0 mA but 30s of 2 mA at the start and the end of the session
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early relapse (2-week follow-up) (Sham Comparator): We compare 5 sessions of active tDCS (2 mA) vs. 5 sessions of sham tDCS (0 mA) to observe if tDCS can reduce early relapse (2-week follow-up). The tDCS is applied during 20 minutes while the patient is watching a documentary about nature. For both active and sham tDCS there is 15-second ramping up and down.
  Interventions: Device: tDCS
- Craving (Experimental): We compare scored craving before and after 5 sessions of either active (2mA) or sham (0mA) tDCS. The tDCS is applied during 20 minutes while the patient is watching a documentary about nature. For both active and sham tDCS there is 15-second ramping up and down.
  Interventions: Device: tDCS
- Working memory (Experimental): We compare reverse memory span before and after 5 sessions of either active (2mA) or sham (0mA) tDCS. The tDCS is applied during 20 minutes while the patient is watching a documentary about nature. For both active and sham tDCS there is 15-second ramping up and down.
  Interventions: Device: tDCS
- Depressive symptoms (Experimental): We compare scored BDI-II before and after 5 sessions of either active (2mA) or sham (0mA) tDCS. The tDCS is applied during 20 minutes while the patient is watching a documentary about nature. For both active and sham tDCS there is 15-second ramping up and down.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — 5 sessions of 20-minute tDCS at 2 mA over the dorsolateral prefrontal cortex (35cm² sponge)

SUMMARY:
Despite the system of care in place, patients suffering from an alcohol use disorder (AUD) continue to relapse after their detoxification. For about twenty years, neuromodulations and their mechanisms have been investigated in research in order to apply it as a therapeutic means, in particular direct current transcranial stimulation (tDCS). A previous study found a reduction of relapse rate thanks to the tDCS over the dorsolateral prefrontal cortex (DLPFC; anode on the right and cathode on the left) combined with an ICT.

This clinical trial of 5 sessions of tDCS alone on the DLPFC (20 minutes, anode on the right, cathode on the left). This study follows the same tDCS configuration as the previous one and takes place in the same multidisciplinary detoxification framework in order to see the relevance of using combined tDCS or only tDCS in clinical practice.

DETAILED DESCRIPTION:
Hypotheses: For patients with AUD five sessions of tDCS during a detoxification:

* decrease the relapse rate 2 weeks after the treatment;
* decrease patient craving;
* decrease depression and anxiety symptoms;
* strengthen working memory performances.

Context: This is a clinical trial that is part of an alcohol detoxification cure at Unit 72 Addictology of CHU Brugmann. The idea is to add a neuromodulation intervention to the initial management, multidisciplinary and psycho-bio-social. This will be a randomized, sham-controlled, single-blind study.

A total of 60 subjects will be recruited according to the inclusion and exclusion criteria. They will be randomly divided into two groups: the 'active' group (A) that will benefit from tDCS stimulation and the 'sham' group (S).

Measures:

Primary dependent variables :

Relapse and total abstinence measured at several defined times: two weeks, one month, three months, six months and one year after treatment.

Secondary dependent variables:

* Craving measured before and after each tDCS session via visual analog scales, such as Likert 0 to 10. Craving will also be measured in T1 and T2 through the Craving Experience Questionnaire (CEQ);
* Symptoms of depression with the Beck Depression Inventory (BDI-II) and positive and negative affectivity with the Positive and Negative Affect Schedule (PANAS) measured at T1 and T2;
* Anxiety trait in T1 and T2 with the State Anxiety Inventory (STAI-A).
* The working memory performance measured in T1 and T2 with the span reversed.

All the questionnaires were in French version.

Metacognition items: At the end of the experiment, patients will be asked orally (1) Do you think you are in the active tDCS group?, (2) Would you be interested in continuing this intervention over a longer period of time?

Statistical analyses:

Primary measurement: In order to respond to our primary assumptions about relapse, a logistic regressions will be performed with the independent variable conditions (tDCS active scored 1 and tDCS sham scored -1) and the variable dependent relapse at each measurement (2 weeks, 1 month, 3 months, 6 months and 1 year). A Kaplan-Meier survival analysis will be performed on the number of days prior to relapse to compare the curves up to one year of follow-up.

Secondary measures: In order to respond to our secondary assumptions about the variables before and after the intervention, mixed repeated measures ANOVAs [Time (T1 vs. T2) x Condition (tDCS active vs. tDCS sham)] will be performed.

ELIGIBILITY:
Inclusion Criteria:

* French speaker
* Severe Alcohol Use Disorder requiring alcohol rehabilitation
* Desire to stay sober for at least the next six months

Exclusion Criteria:

* Neurological history (epilepsy, head injury, and stroke)
* Mental confusion or severe cognitive impairment
* Schizophrenia, chronic psychotic disorders or bipolar type 1 disorder
* Metal in the brain
* Pregnancy
* Having participated in our previous study combining tDCS with ICT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Relapse rate 2 weeks after discharge | 2-week follow-up
  by phone call; more than 60 g of alcohol
Relapse rate 1 month after discharge | 1-month follow-up
  by phone call; more than 60 g of alcohol
Relapse rate 3 months after discharge | 3-month follow-up
  by phone call; more than 60 g of alcohol

SECONDARY OUTCOMES:
Craving | at pre-intervention (day 12 of hospitalization)
  Visual Analog Scales (4 items, range 1-9 each; 1 = no craving, 9 = extreme craving)
Craving | at post-intervention (day 22 of hospitalization)
  Visual Analog Scales (4 items, range 1-9 each; 1 = no craving, 9 = extreme craving)
Working memory | at pre-intervention (day 12 of hospitalization)
  Reverse memory span, range 2-9
Working memory | at post-intervention (day 22 of hospitalization)
  Reverse memory span, range 2-9
Depressive symptoms | at pre-intervention (day 12 of hospitalization)
  Beck Depression Inventory II (BDI-II) [44], which assessed the severity of depressive symptoms (21 items; range, 0-63; 10-18 = mild depression, 19-29 = moderate depression, 30-63 = severe depression)
Depressive symptoms | at post-intervention (day 22 of hospitalization)
  Beck Depression Inventory II (BDI-II) [44], which assessed the severity of depressive symptoms (21 items; range, 0-63; 10-18 = mild depression, 19-29 = moderate depression, 30-63 = severe depression)
Anxiety state | at pre-intervention (day 12 of hospitalization)
  The State-Trait Anxiety Inventory (STAI-Y) A which assessed the anxiety state (20 items; range, 20-80; < 35 = very low anxiety state, 36-45 = low anxiety state, 46-55 = medium anxiety state, 56-65 = high anxiety state, >65 = very high anxiety state).
Anxiety state | at post-intervention (day 22 of hospitalization)
  The State-Trait Anxiety Inventory (STAI-Y) A which assessed the anxiety state (20 items; range, 20-80; < 35 = very low anxiety state, 36-45 = low anxiety state, 46-55 = medium anxiety state, 56-65 = high anxiety state, >65 = very high anxiety state).

CONTACTS AND LOCATIONS:
Overall Officials: Dubuson Macha, MA, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- CHU-Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT04990375/Prot_SAP_000.pdf